CLINICAL TRIAL: NCT00004635
Title: A Double Blinded Randomized Crossover Phase III Study of Oral Thalidomide Versus Placebo in Patients With Stage D0 Androgen Dependent Prostate Cancer Following Limited Hormonal Ablation
Brief Title: Thalidomide for the Treatment of Hormone-Dependent Prostate Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Collaborators: Holy Cross Hospital, Fort Lauderdale (Unknown); Louisiana State University Health Sciences Center in New Orleans (Other); Wayne State University (Other); University of Minnesota (Other); Columbia University (Other); University of Pittsburgh (Other); United States Naval Medical Center, Portsmouth (U.S. Federal Agency); University of Washington (Other)
Responsible Party: Principal Investigator, William Dahut Jr., M.D., Principal Investigator, National Institutes of Health Clinical Center (CC)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 000080; 00-C-0080 (Other: Clinical Center, NIH); 000080 (Other: Clinical Center, NIH); NCT00020085 (obsolete NCT alias)
Record Dates: First submitted 2000-02-19; First posted 2000-02-21 (Estimated); Results first posted 2012-09-12 (Estimated); Last update posted 2018-05-22 (Actual); Status verified 2018-04

CONDITIONS: Prostate Cancer
Keywords: Angiogenesis; Cancer; Hormonal Therapy; Prostate; Thalidomide; Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms; Neoplasms | interventions — Thalidomide; Leuprolide; Goserelin; Sugars

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Thalidomide (Experimental): Study participants are randomly assigned to one of two treatment groups. Participants received leuprolide or goserelin for 6 months. In period 1 participants received thalidomide orally 200 mg a day. Patients will be followed until PSA progression defined as prostate-specific antigen (PSA) level that returns to what it was before beginning leuprolide or goserelin or to 5 nanograms per liter, whichever is lower. The participants are returned to the leuprolide or goserelin treatment for 6 months. In period 2 participants received the placebo for thalidomide once a day.
  Interventions: Drug: Thalidomide; Drug: leuprolide acetate; Drug: goserelin
- Placebo (Experimental): Study participants are randomly assigned to one of two treatment groups. Participants received leuprolide or goserelin for 6 months. In period 1 participants received placebo for thalidomide. Patients will be followed until PSA progression defined as prostate-specific antigen (PSA) level that returns to what it was before beginning leuprolide or goserelin or to 5 nanograms per liter, whichever is lower. The participants are returned to the leuprolide or goserelin treatment for 6 months. In period 2 participants received thalidomide 200 mg once a day.
  Interventions: Drug: leuprolide acetate; Drug: goserelin; Other: Placebo

INTERVENTIONS:
Drug: Thalidomide — Thalidomide 200 mg given orally every evening at 9pm. Treatment may continue indefinitely provided that there are no dose-limiting toxicity.
  Other Names: Thalomid
  Arms: Thalidomide
Drug: leuprolide acetate — Injections of leuprolide once a month for six months.
  Other Names: leuprorelin
Drug: goserelin — Injections of Goserelin once a month for six months.
  Other Names: Zolodex
Other: Placebo — Patients will receive the placebo if they initially received thalidomide. The starting dose of placebo 200 mg (four capsules of 100-50 mg capsules) orally once daily at bedtime.
  Other Names: Sugar pill
  Arms: Placebo

SUMMARY:
This multi-center study will evaluate whether thalidomide can improve the effectiveness of the drugs leuprolide or goserelin in treating testosterone-dependent prostate cancer. Leuprolide and goserelin-both approved to treat prostate cancer-reduce testosterone production, which, in most patients, reduces the size of the tumor. Thalidomide, a drug used for many years to treat leprosy, blocks the growth of blood vessels that may be important to disease progression.

Patients 18 years or older with testosterone-dependent prostate cancer that has persisted or recurred after having had surgery, radiation therapy, or cryosurgery, but whose disease has not metastasized (spread beyond the prostate) may be eligible for this study. Candidates are screened with a medical history and physical examination, including blood tests, bone and computed tomography (CT) scans or other imaging studies.

Study participants are randomly assigned to one of two treatment groups. One group receives leuprolide or goserelin followed by thalidomide; the other receives leuprolide or goserelin followed by placebo (a look-alike pill with no active ingredients). Patients in both groups receive an injection of leuprolide or goserelin once a month for 6 months. After that time they take four capsules of either thalidomide or placebo once a day and remain on the drug until their prostate-specific antigen (PSA) level returns to what it was before beginning leuprolide or goserelin or to 5 nanograms per liter, whichever is lower.(PSA is a protein secreted by the prostate gland. Monitoring changes in levels of this protein can help evaluate tumor progression). At this point the entire procedure begins again, starting with leuprolide or goserelin treatment, but the experimental drug is switched; patients originally treated with thalidomide are crossed over to placebo, and patients originally treated with placebo are crossed over to thalidomide.

Patients are monitored periodically with the following tests and procedures:

Medical histories and physical examinations. Blood and urine tests to monitor thalidomide and PSA levels, the response to treatment, and routine laboratory values (e.g., cell counts and kidney and liver function).

Computed tomography (CT) and bone scans, and possibly other imaging tests to assess the tumor.

Electromyography (EMG) and nerve conduction studies, as needed. For electromyography, a thin needle is inserted into a few muscles and the patient is asked to relax or to contract the muscles.

DETAILED DESCRIPTION:
This is a double-blind randomized phase III study designed to determine if thalidomide can improve the efficacy of the luteinizing hormone releasing hormone (LHRH) agonist (leuprolide or goserelin) in hormone-responsive patients with a rising PSA after primary definitive therapy for prostate cancer. Patients with only a rising PSA will be randomized to LHRH agonist for six months followed by oral thalidomide 200 mg per day or placebo (phase A). At the time of PSA progression, an LHRH agonist will be restarted for six additional months. After six months, patients originally treated with thalidomide will be crossed over to placebo and patients originally treated with placebo will be crossed over to thalidomide and followed until PSA progression or the development of metastatic disease, whichever occurs first (Phase B). Additional information will be obtained on changes in the circulating levels of the following growth factors: basic fibroblast growth factor (bFGF), tumor necrosis factor (TNF), vascular endothelial growth factor (VEGF), and transforming growth factor beta (TGFbeta). Likewise we will monitor changes in testosterone and dihydrotestosterone (DHT) throughout the study. Neurological complications are the primary dose-limiting toxicity anticipated with chronic thalidomide administration.

ELIGIBILITY:
* Inclusion Criteria:
* patients must have prostate specific antigen (PSA) only androgen dependent adenocarcinoma of the prostate. All patients must have failed definitive therapy (radical prostatectomy, radiation therapy with external beam or brachytherapy,or cryosurgery).
* Patients must have a negative Computerized Tomography (CT) scan and Bone Scan for metastatic prostate cancer.
* Patients must have histopathological documentation of prostate cancer. Every attempt should be made to have slides and blocks reviewed at National Cancer Institute (NCI) Pathology laboratory. The review of pathology by the NCI will not delay enrollment.
* Patients must have progressive prostate cancer. Two consecutively rising PSAs above the nadir post-definitive therapy and an absolute value greater than 1.0 ng/ml separated by at least 2 weeks.
* Patients must have a life expectancy of more than 12 months.
* Patients must have a performance status of 0 to 2 according to the Eastern Cooperative Oncology Group (ECOG) criteria.
* Hematological eligibility parameters (within 2 weeks of starting therapy):

Granulocyte count greater than or equal to 1,000/mm^3. Platelet count greater than or equal to 75,000/mm^3.

- Biochemical eligibility parameters (within 2 weeks of starting therapy): If the creatinine is greater than 2.0 mg/dL obtain a 24 hour urine collection.

Creatinine clearance must be greater than 40 mL/min. Hepatic function:

bilirubin (total) less than or equal to 1 mg/dL upper limit of normal; Alanine aminotransferase (ALT) less than 2.5 times upper limit of normal.

* Exception: Patients with Clinical Gilbert's Syndrome may have total bilirubin less than or equal to 2.5 mg/dL.
* Patients must not have other concurrent malignancies (within the past 2 years) with the exception of nonmelanoma skin cancer and Rai Stage 0 chronic lymphoma leukemia), in situ carcinoma of any site, or life threatening illnesses, including untreated infection (must be at least 1 week off intravenous antibiotic therapy before beginning thalidomide).
* Patients with a history of unstable or newly diagnosed angina pectoris, recent myocardial infarction (within 6 months of enrollment), New York class II-IV congestive heart failure, chronic obstructive lung disease requiring oxygen therapy, uncontrolled seizure activity or by medical judgement of the physician, are not eligible.
* Patients must be able to understand and sign an informed consent document.
* Patients must be willing to travel from their home to the NIH or the participating institution (Louisiana State Univ., Univ. of Washington, Columbia University,Wayne State, University of Minnesota, University of Pittsburgh, Holy Cross)for follow-up visits (due to sedation associated with thalidomide). It is preferred that patients not drive the first 3 days of taking daily dosing,or if sedation appears to be a continuing complication).
* Patients must be greater than or equal to 18 years of age.
* Male patients must be counseled about the possibility that thalidomide may be present in semen. Men must use a latex condom every time they have sexual intercourse with women during therapy and for 8 weeks after discontinuing thalidomide, even if they have had a successful vasectomy.
* Patients may enroll as a late entry if the following criteria are met: Have received leuprolide or goserelin within 3 months of starting study,have a PSA within two weeks of hormonal injection and have a bone scan without metastasis within 8 weeks of enrollment.
* Patients with Rai Stage of Chronic Lymphocytic Leukemia (lymphocytosis only) will be eligible.
* Exclusion Criteria:
* Patients that have received leuprolide, diethylstilbestrol (DES), flutamide, bicalutamide, PC stands for prostate cancer and SPES is the Latin word for hope)PC-SPES, goserelin, cytotoxic chemotherapy, finasteride and/or nilutamide within the past year (or currently) are not eligible. Patients that received these agents for adjuvant or neoadjuvant therapy at the time of definitive therapy are eligible. Exception: Patients enrolled under late entry criteria, who have received leuprolide/goserelin within 3 months of starting study are eligible.
* Patients with National Cancer Institute (NCI)/Cancer Therapy Evaluation Program (CTEP) grade 2 or greater peripheral neuropathy of any cause that is clinically detectable, patients receiving anti-convulsive medications, and patients with a history of seizures within the past 10 years will not be eligible for this study.
* Patients who are receiving sedative/hypnotic agents (i.e. benzodiazepines) which cannot be discontinued, will not be eligible for this study. Patients who have had a surgical orchiectomy will not be eligible for this study.
* Patients who received a systemic chemotherapy for prostate cancer will not be eligible.
* Patients with a confirmed psychiatric history of a major depression consistent with American Psychiatric Association Diagnostic and Statistical Manual (DSM IIIR criteria), confirmed by a psychiatrist will not be eligible.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 159 (Actual)
Dates: Start 2000-03-01 (Actual); Primary Completion 2005-01-30 (Actual); Study Completion 2010-03-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William L Dahut, M.D., Principal Investigator — National Cancer Institute, National Institutes of Heath
Locations (9):
- United States (9):
  - Holy Cross Hospital, Fort Lauderdale, Fort Lauderdale, Florida
  - Louisiana State University, New Orleans, Louisiana
  - National Institutes of Health, Clinical Center, 9000 Rockville Pike, Bethesda, Maryland
  - Wayne State University Hutzel Hospital, Detroit, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - Columbia University, New York, New York
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Naval Medical Center, Portsmouth, Portsmouth, Virginia
  - University of Washington, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Aronson IK, Yu R, West DP, Van den Broek H, Antel J. Thalidomide-induced peripheral neuropathy. Effect of serum factor on nerve cultures. Arch Dermatol. 1984 Nov;120(11):1466-70. doi: 10.1001/archderm.120.11.1466. PMID 6093713
- [Background] Bakay B, Nyhan WL. Binding of thalidomide by macromolecules in the fetal and maternal rat. J Pharmacol Exp Ther. 1968 Jun;161(2):348-60. No abstract available. PMID 5652850
- [Background] Bauer KS, Dixon SC, Figg WD. Inhibition of angiogenesis by thalidomide requires metabolic activation, which is species-dependent. Biochem Pharmacol. 1998 Jun 1;55(11):1827-34. doi: 10.1016/s0006-2952(98)00046-x. PMID 9714301
- [Result] Figg WD, Hussain MH, Gulley JL, Arlen PM, Aragon-Ching JB, Petrylak DP, Higano CS, Steinberg SM, Chatta GS, Parnes H, Wright JJ, Sartor O, Dahut WL. A double-blind randomized crossover study of oral thalidomide versus placebo for androgen dependent prostate cancer treated with intermittent androgen ablation. J Urol. 2009 Mar;181(3):1104-13; discussion 1113. doi: 10.1016/j.juro.2008.11.026. Epub 2009 Jan 23. PMID 19167733
- [Derived] Hawley JE, Pan S, Figg WD, Lopez-Bujanda ZA, Strope JD, Aggen DH, Dallos MC, Lim EA, Stein MN, Hu J, Drake CG. Association between immunosuppressive cytokines and PSA progression in biochemically recurrent prostate cancer treated with intermittent hormonal therapy. Prostate. 2020 Mar;80(4):336-344. doi: 10.1002/pros.23948. Epub 2020 Jan 3. PMID 31899823
- See also: MedlinePlus — http://www.nlm.nih.gov/medlineplus
- See also: Drug Information Portal — http://druginfo.nlm.nih.gov/drugportal/drugportal.jsp
- See also: U.S. FDA Resources — http://www.clinicaltrials.gov/ct2/info/fdalinks

RESULTS

PARTICIPANT FLOW:
Recruitment Details: With nine institutions participating (NCI intramural, Columbia in NY, LSU in New Orleans, Wayne State Univ., Univ. of Washington, Univ. of Minnesota, Univ. of Pittsburgh, Holy Cross and Portsmouth Naval Hosp.)it is expected that 16 pts per mo (190 per year) can be entered onto the trial with an estimated completion of accrual expected in 18 months.
Pre-assignment Details: While patients are crossed-over to the other therapy, because the time until crossover is dependent on time until progression, this differs from a classic crossover study in which patients are followed on both arms for a fixed period of time, evaluated, given a wash-out period, and then followed identically on the other agent.
Groups:
- Thalidomide Followed by Placebo: Study participants are randomly assigned to one of two treatment groups. Participants received leuprolide or goserelin for 6 months. In period 1 participants received thalidomide orally 200 mg a day. Patients will be followed until PSA progression defined as prostate-specific antigen (PSA) level that returns to what it was before beginning leuprolide or goserelin or to 5 nanograms per liter, whichever is lower. The participants are returned to the leuprolide or goserelin treatment for 6 months. In period 2 participants received the placebo for thalidomide once a day.
- Placebo Followed by Thalidomide: Study participants are randomly assigned to one of two treatment groups. Participants received leuprolide or goserelin for 6 months. In period 1 participants received placebo for thalidomide. Patients will be followed until PSA progression defined as prostate-specific antigen (PSA) level that returns to what it was before beginning leuprolide or goserelin or to 5 nanograms per liter, whichever is lower. The participants are returned to the leuprolide or goserelin treatment for 6 months. In period 2 participants received thalidomide 200 mg once a day.
Period: Period One
Arm/Group | Thalidomide Followed by Placebo | Placebo Followed by Thalidomide
Started | 79 | 80
Received Treatment | 73 | 75
Completed | 73 | 74
Not Completed | 6 | 6
Not completed — refused | 2 | 1
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Protocol Violation | 1 | 0
Not completed — PSA did not go <5 ng/mL | 1 | 0
Not completed — second malignancy | 1 | 0
Not completed — progressed | 0 | 2
Not completed — health problem | 0 | 1
Not completed — discrepancy in data entry | 0 | 1
Period: Period Two
Arm/Group | Thalidomide Followed by Placebo | Placebo Followed by Thalidomide
Started | 44 | 59
Completed | 38 | 50
Not Completed | 6 | 9
Not completed — progression | 2 | 3
Not completed — Adverse Event | 1 | 0
Not completed — refused | 0 | 2
Not completed — health problem | 1 | 1
Not completed — travel issues | 0 | 1
Not completed — secondary malignancy | 1 | 1
Not completed — Lost to Follow-up | 1 | 0
Not completed — discrepancy in data entry | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Thalidomide Followed by Placebo | Placebo Followed by Thalidomide | Total
Number analyzed (Participants) | 79 | 80 | 159
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 41 | 28 | 69
  >=65 years | 38 | 52 | 90
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.35 (7.43) | 68.46 (8.54) | 66.91 (7.98)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 79 | 80 | 159
Region of Enrollment [Number; unit: participants]
  United States | 79 | 80 | 159

OUTCOME MEASURES:

1. Primary Outcome: Time to Progression
Description: Time to progression is defined as follows: if the PSA returns to baseline (defined as the PSA value prior to starting leuprolide or goserelin) or increases to the absolute value of 5 ng/ml.
Time Frame: 36 months
Population: Per protocol. First intervention phase-73 participants (thalidomide) were analyzed and 0 was excluded; 74 participants were analyzed (placebo) and 1 was excluded for discrepancy in data entry. Crossover phase-50 participants were analyzed (thalidomide)and 1 was excluded for discrepancy in data entry, 38 participants for placebo and 0 excluded.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Thalidomide: Participants who received thalidomide in period 1 or 2.
- Placebo: Participants who received placebo in period 1 or 2
Arm/Group | Thalidomide | Placebo
Number analyzed (Participants) | 123 | 112
months | 15 [12.0 to 22.1] | 9.6 [8.5 to 12.9]

2. Secondary Outcome: The Number of Participants With Adverse Events
Description: Here are the total number of participants with adverse events. For the detailed list of adverse events see the adverse event module.
Time Frame: Date treatment consent signed to date off study, approximately 60 months
Measure: Count of Participants; unit: Participants
Arm/Group | Thalidomide | Placebo
Number analyzed (Participants) | 138 | 124
Participants | 117 | 98

ADVERSE EVENTS:
Time Frame: Date treatment consent signed to date off study, approximately 5 years.
Arm/Group | Thalidomide | Placebo | Goserelin (Zoladex) | Leuprolide
All-Cause Mortality (participants affected / at risk) | 0/138 | 0/124 | 0/159 | 0/159
Serious Adverse Events (participants affected / at risk) | 117/138 | 98/124 | 13/159 | 124/159
Other Adverse Events (participants affected / at risk) | 67/138 | 63/124 | 10/159 | 66/159
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Thalidomide (N=138) | Placebo (N=124) | Goserelin (Zoladex) (N=159) | Leuprolide (N=159)
Allergic reaction/hypersensitivity (including drug fever) (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain or cramping (Reproductive system and breast disorders) | 5 (5) | 2 (2) | 0 (0) | 0 (0)
Alkaline phosphatase (Investigations) | 2 (2) | 4 (5) | 0 (0) | 4 (4)
Allergic rhinitis (including sneezing, nasal stuffiness, postnasal drip) (Immune system disorders) | 3 (3) | 2 (2) | 0 (0) | 1 (1)
Chest pain (non-cardiac and non-pleuritis) (General disorders) | 5 (5) | 1 (1) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 5 (5) | 1 (1) | 0 (0) | 0 (0)
Anorexia (Gastrointestinal disorders) | 3 (4) | 0 (0) | 0 (0) | 1 (1)
Arrhythmia-other (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (joint pain) (Musculoskeletal and connective tissue disorders) | 5 (5) | 5 (5) | 0 (0) | 3 (4)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Ataxia (incoordination) (Nervous system disorders) | 12 (14) | 1 (1) | 0 (0) | 1 (1)
Bilirubin (Investigations) | 8 (11) | 16 (22) | 0 (0) | 4 (4)
Brusing (in absence of grade 3 or 4 thrombocytopenia) (Blood and lymphatic system disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
CNS cerebrovascular ischemia (Nervous system disorders) | 3 (3) | 1 (1) | 0 (0) | 1 (1)
CPK (creatine phosphokinase) (Investigations) | 4 (5) | 5 (5) | 0 (0) | 1 (1)
Circulatory or cardiac-Other (Cardiac disorders) | 3 (3) | 2 (2) | 0 (0) | 0 (0)
Cognitive disturbance/learning problems (Nervous system disorders) | 3 (5) | 0 (0) | 0 (0) | 0 (0)
Confusion (Psychiatric disorders) | 8 (8) | 2 (3) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 85 (116) | 32 (42) | 1 (1) | 3 (3)
Bone pain (Musculoskeletal and connective tissue disorders) | 5 (7) | 1 (1) | 0 (0) | 0 (0)
Constitutional symptoms-Other (General disorders) | 2 (4) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 8 (8) | 0 (0) | 1 (1)
Creatinine (Investigations) | 4 (5) | 4 (5) | 0 (0) | 4 (4)
Depressed level of consciousness (Nervous system disorders) | 33 (38) | 5 (5) | 0 (0) | 2 (2)
Derma/Skin-Other: Lower lip lesion (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diarrhea (without colostomy) (Gastrointestinal disorders) | 8 (8) | 8 (8) | 0 (0) | 3 (3)
Dizziness/lightheadedness (Nervous system disorders) | 58 (67) | 18 (22) | 0 (0) | 2 (2)
Dry eye (Eye disorders) | 6 (6) | 2 (2) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 17 (19) | 5 (5) | 0 (0) | 0 (0)
Dyspepsia/heartburn (Gastrointestinal disorders) | 4 (4) | 5 (5) | 0 (0) | 0 (0)
Dysphagia, esophagitis, odynophagia (painful swallowing) (Gastrointestinal disorders) | 2 (3) | 1 (1) | 0 (0) | 0 (0)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 36 (42) | 13 (16) | 0 (0) | 2 (2)
Dysuria (painful urination) (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Edema (General disorders) | 39 (50) | 11 (13) | 0 (0) | 3 (3)
Erectile impotence (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 1 (1) | 11 (11)
Extrapyramidal/involuntary movement/restlessness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Fatigue (lethargy, malaise, asthenia) (General disorders) | 66 (91) | 37 (47) | 4 (5) | 21 (22)
Fever (in absence of neutropenia, where neutropenia is defined as AGC<1.0x109/L) (General disorders) | 1 (2) | 0 (0) | 0 (0) | 1 (2)
Flatulence (Gastrointestinal disorders) | 1 (1) | 4 (4) | 0 (0) | 0 (0)
Flushing (Vascular disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
GI-Other (Gastrointestinal disorders) | 4 (4) | 3 (4) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Gynecomastia (Reproductive system and breast disorders) | 7 (7) | 4 (4) | 1 (1) | 3 (3)
Headache (Nervous system disorders) | 25 (28) | 13 (13) | 0 (0) | 4 (5)
Hearing-Other (Ear and labyrinth disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Hematologic-Other (Blood and lymphatic system disorders) | 1 (1) | 3 (5) | 0 (0) | 5 (5)
Hematuria (in the absence of vaginal bleeding) (Renal and urinary disorders) | 2 (2) | 2 (2) | 0 (0) | 1 (1)
Hemoglobin (Hgb) (Investigations) | 21 (25) | 8 (13) | 0 (0) | 8 (8)
Hemolysis (e.g., immune hemolytic anemia, drug-related hemolysis, other (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hiccoughs (hiccups, singultus) (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hot flashes/flashes (Vascular disorders) | 11 (11) | 9 (13) | 11 (13) | 102 (130)
Hypercalcemia (Metabolism and nutrition disorders) | 3 (3) | 3 (3) | 0 (0) | 3 (3)
Hyperglycemia (Metabolism and nutrition disorders) | 30 (48) | 24 (27) | 0 (0) | 10 (11)
Hyperkalemia (Metabolism and nutrition disorders) | 4 (9) | 6 (8) | 0 (0) | 1 (1)
Hypermagnesemia (Metabolism and nutrition disorders) | 2 (3) | 4 (4) | 0 (0) | 3 (3)
Hypernatremia (Metabolism and nutrition disorders) | 4 (4) | 3 (3) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 5 (6) | 0 (0) | 0 (0) | 2 (2)
Hypoalbuminemia (Metabolism and nutrition disorders) | 24 (30) | 15 (26) | 0 (0) | 9 (9)
Hypoglycemia (Metabolism and nutrition disorders) | 2 (3) | 4 (6) | 0 (0) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Hypomagnesmia (Metabolism and nutrition disorders) | 15 (16) | 4 (4) | 0 (0) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 4 (4) | 3 (4) | 0 (0) | 1 (1)
Hypophosphatemia (Metabolism and nutrition disorders) | 5 (7) | 3 (4) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 9 (9) | 4 (4) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Incontinence (Renal and urinary disorders) | 7 (7) | 2 (2) | 0 (0) | 2 (2)
Infection without neutropenia (Infections and infestations) | 8 (13) | 9 (14) | 0 (0) | 1 (2)
Infection, Other (Infections and infestations) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Inner ear/hearing (Ear and labyrinth disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 11 (12) | 1 (1) | 5 (6)
Joint, muscle, or bone (osseous)-Other (Musculoskeletal and connective tissue disorders) | 6 (7) | 4 (9) | 1 (1) | 0 (0)
Leukocytes (total WBC) (Investigations) | 13 (23) | 4 (19) | 0 (0) | 2 (2)
Libido (Psychiatric disorders) | 2 (2) | 0 (0) | 1 (1) | 13 (14)
Lymphatics (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 7 (12) | 4 (5) | 0 (0) | 1 (1)
Memory loss (Nervous system disorders) | 9 (9) | 3 (3) | 0 (0) | 0 (0)
Mood alteration-anxiety agitation (Psychiatric disorders) | 11 (12) | 3 (3) | 0 (0) | 1 (1)
Mood alteration-depression (Psychiatric disorders) | 11 (11) | 5 (5) | 0 (0) | 3 (3)
Mouth dryness (Gastrointestinal disorders) | 44 (45) | 13 (15) | 0 (0) | 0 (0)
Muscle cramps (thigh) (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Muscle weakness (not due to neuropathy) (Musculoskeletal and connective tissue disorders) | 10 (11) | 1 (1) | 1 (1) | 1 (1)
Myalgia (muscle ache) (Musculoskeletal and connective tissue disorders) | 20 (20) | 11 (13) | 0 (0) | 4 (4)
Nail changes (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 15 (20) | 10 (11) | 0 (0) | 1 (1)
Neurologic-Other (Nervous system disorders) | 7 (8) | 2 (2) | 0 (0) | 1 (1)
Neuropathy cranial (Nervous system disorders) | 4 (6) | 0 (0) | 0 (0) | 0 (0)
Neuropathy motor (Nervous system disorders) | 8 (9) | 1 (1) | 0 (0) | 0 (0)
Neuropathy-sensory (Nervous system disorders) | 55 (93) | 23 (31) | 0 (0) | 6 (6)
Neutrophils/granulocytes (ANC/AGC) (Investigations) | 9 (18) | 4 (9) | 0 (0) | 0 (0)
Ocular-Other (Eye disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Pain-Other (Nervous system disorders) | 5 (5) | 6 (8) | 0 (0) | 4 (4)
Palpitation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Petechiae/purpura (hemorrhage/bleeding into skin or mucosa) (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Photosensitivity (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Platelets (Investigations) | 3 (3) | 4 (6) | 0 (0) | 3 (3)
Protrombin Time/INR-International Normalized Ratio of protrombin time (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (4) | 0 (0) | 1 (1)
Pulmonary-Other (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 2 (2) | 0 (0) | 1 (1)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 26 (30) | 14 (16) | 0 (0) | 3 (3)
Rectal bleeding/hematochezia (Gastrointestinal disorders) | 1 (1) | 6 (7) | 0 (0) | 1 (1)
Rectal or perirectal pain (proctalgia) (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
SGOT (AST) (Investigations) | 10 (12) | 16 (23) | 0 (0) | 12 (14)
SGPT (ALT) (Investigations) | 9 (11) | 12 (16) | 0 (0) | 16 (18)
Salivary gland changes (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Secondary Malignancy-Other (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Sense of smell (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 28 (31) | 5 (5) | 0 (0) | 1 (1)
Skin-Other (Skin and subcutaneous tissue disorders) | 3 (3) | 5 (5) | 0 (0) | 1 (1)
Stomatitis/pharyngitis (oral/pharyngeal mucositis) (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Supraventricular arrhythmias (SVT/atrial fibrillation/flutter) (Cardiac disorders) | 2 (2) | 2 (3) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 4 (6) | 0 (0) | 0 (0) | 0 (0)
Taste disturbance (dysgeusia) (Gastrointestinal disorders) | 4 (4) | 3 (3) | 0 (0) | 0 (0)
Tearing (watery eyes) (Eye disorders) | 3 (3) | 0 (0) | 0 (0) | 1 (2)
Thrombosis/embolism (Vascular disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (1)
Tremor (Nervous system disorders) | 18 (19) | 3 (4) | 0 (0) | 0 (0)
Urinary frequency/urgency (Renal and urinary disorders) | 2 (3) | 4 (4) | 1 (1) | 8 (8)
Urticaria (hives, welts, wheals) (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Ventricular arrhythmia (PVCs/bigeminy/trigeminy/ventricular tachycardia) (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vision-blurred vision (Eye disorders) | 8 (9) | 3 (3) | 0 (0) | 1 (1)
Vision-double vision (diplopia) (Eye disorders) | 1 (1) | 2 (3) | 0 (0) | 0 (0)
Vision-flashing lights/floaters (Eye disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Vision-night blindness (nyctalopia) (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Voice changes/stridor/larynx (e.g., hoarsneness, loss of voice, laryngitis) (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 4 (4) | 3 (3) | 0 (0) | 0 (0)
Weight gain (Investigations) | 9 (11) | 3 (4) | 0 (0) | 1 (1)
Weight loss (Investigations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Wound-infectious (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Renal/GU-Other (Renal and urinary disorders) | 4 (5) | 4 (5) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Sweating (diaphoresis) (Skin and subcutaneous tissue disorders) | 2 (3) | 0 (0) | 0 (0) | 4 (6)
Cardiac-ischemia/infarction (Cardiac disorders) | 2 (2) | 1 (1) | 0 (0) | 2 (2)
Cardiac-left ventricular function (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Endocrine-Other (Endocrine disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Impotency (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
LDH (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Metabolic-Other (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neuropathic pain (e.g., jaw pain, neurologic pain, phantom limb pain, post-infectious neuralgia, or (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (non-malignant) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rigors/chills (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypercholesterolemia (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vision-photophobia (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Seizure(s) (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vasovagal episode (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 2 (4) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Thalidomide (N=138) | Placebo (N=124) | Goserelin (Zoladex) (N=159) | Leuprolide (N=159)
Allergic rhinitis (including sneezing, nasal stuffiness, postnasal drip) (Immune system disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain or cramping (Reproductive system and breast disorders) | 2 (2) | 3 (3) | 0 (0) | 0 (0)
Alkaline phosphatase (Investigations) | 2 (3) | 1 (1) | 0 (0) | 3 (3)
Bone pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (2) | 0 (0) | 0 (0)
Cardiac left ventricular function (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac-ischemia/infarction (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Cataract (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Circulatory or cardiac-Other (Cardiac disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Endocrine-Other (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Coag-Other (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 2 (2) | 1 (1) | 0 (0)
Creatinine (Investigations) | 9 (11) | 5 (7) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Dizziness/lightheadedness (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 3 (4)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia/heartburn (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (4) | 0 (0) | 1 (1)
Fatigue (lethargy, malaise, asthenia) (General disorders) | 2 (2) | 1 (1) | 1 (2) | 3 (3)
Headache (Nervous system disorders) | 2 (2) | 1 (1) | 0 (0) | 2 (2)
Hearing-Other (Ear and labyrinth disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Hematuria (in the absence of vaginal bleeding) (Renal and urinary disorders) | 1 (1) | 1 (2) | 0 (0) | 1 (1)
Hemoglobin (Hgb) (Blood and lymphatic system disorders) | 3 (3) | 3 (4) | 0 (0) | 6 (8)
Hypercalcemia (Metabolism and nutrition disorders) | 3 (3) | 4 (4) | 0 (0) | 3 (3)
Hyperglycemia (Metabolism and nutrition disorders) | 12 (17) | 13 (23) | 3 (3) | 13 (14)
Hyperkalemia (Metabolism and nutrition disorders) | 4 (4) | 0 (0) | 0 (0) | 1 (2)
Hypermagnesemia (Metabolism and nutrition disorders) | 2 (2) | 2 (2) | 0 (0) | 1 (1)
Hypernatremia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 3 (3) | 3 (3) | 0 (0) | 2 (2)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperuricemia (Metabolism and nutrition disorders) | 2 (4) | 6 (6) | 0 (0) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 8 (10) | 3 (3) | 0 (0) | 2 (2)
Hypoglycemia (Metabolism and nutrition disorders) | 4 (4) | 2 (2) | 0 (0) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hypomagnesmia (Metabolism and nutrition disorders) | 2 (3) | 1 (1) | 0 (0) | 3 (4)
Hyponatremia (Metabolism and nutrition disorders) | 3 (3) | 0 (0) | 0 (0) | 2 (3)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (2) | 1 (2) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Incontinence (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0) | 3 (3)
Infection without neutropenia (Infections and infestations) | 9 (10) | 7 (11) | 0 (0) | 3 (3)
Infection, Other (Infections and infestations) | 1 (1) | 6 (7) | 1 (1) | 0 (0)
Inner ear/hearing (Ear and labyrinth disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Joint, muscle, or bone (osseous)-Other (Musculoskeletal and connective tissue disorders) | 4 (4) | 7 (11) | 2 (2) | 3 (3)
Leukocytes (total WBC) (Investigations) | 2 (2) | 1 (2) | 0 (0) | 1 (1)
Middle ear/hearing (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mood alteration-anxiety agitation (Psychiatric disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Mouth dryness (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (2) | 0 (0)
Myalgia (muscle ache) (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 0 (0) | 2 (2)
Myositis (inflammation/damage of muscle) (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neuropathic pain (e.g., jaw pain, neurologic pain, phantom limb pain, post-infectious neuralgia, or (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neuropathy-sensory (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Neutrophils/granulocytes (ANC/AGC) (Investigations) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Ocular-Other (Ear and labyrinth disorders) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
Pain-Other (Nervous system disorders) | 3 (3) | 10 (12) | 2 (3) | 3 (3)
Photosensitivity (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Platelets (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Pulmonary-Other (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 7 (7) | 2 (4) | 1 (1) | 1 (1)
Renal/GU-Other (Renal and urinary disorders) | 1 (1) | 3 (5) | 0 (0) | 0 (0)
SGPT (ALT) (Investigations) | 1 (1) | 0 (0) | 0 (0) | 3 (3)
Secondary Malignancy-Other (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1) | 0 (0) | 3 (3)
Sinus bradycardia (Cardiac disorders) | 2 (3) | 3 (3) | 0 (0) | 2 (2)
Skin-Other (Skin and subcutaneous tissue disorders) | 3 (4) | 3 (5) | 2 (2) | 1 (1)
Stomatitis/pharyngitis (oral/pharyngeal mucositis) (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Trauma R. big toe (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ureteral obstruction (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary frequency/urgency (Renal and urinary disorders) | 2 (3) | 4 (4) | 1 (1) | 0 (0)
Voice changes/stridor/larynx (e.g., hoarsneness, loss of voice, laryngitis) (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Wound (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (joint pain) (Musculoskeletal and connective tissue disorders) | 0 (0) | 6 (6) | 0 (0) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
CPK (creatine phosphokinase) (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (2)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Diarrhea (without colostomy) (Gastrointestinal disorders) | 0 (0) | 3 (3) | 0 (0) | 1 (1)
Edema (General disorders) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Erectile impotence (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hematologic-Other (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hepatic-Other (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hot flashes/flashes (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Hypocalcemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Infection with unknown ANC (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Insomnia (Psychiatric disorders) | 0 (0) | 3 (3) | 0 (0) | 1 (1)
Mood alteration-depression (Psychiatric disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Proctitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rectal bleeding/hematochezia (Gastrointestinal disorders) | 0 (0) | 6 (6) | 0 (0) | 2 (2)
SGOT (AST) (Investigations) | 0 (0) | 2 (3) | 0 (0) | 1 (1)
Supraventricular arrhythmias (SVT/atrial fibrillation/flutter) (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Taste disturbance (dysgeusia) (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Weight loss (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sweating (diaphoresis) (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1) | 2 (2)
Muscle weakness (not due to neuropathy) (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
GI-Other (Gastrointestinal disorders) | 0 (0) | 1 (3) | 1 (2) | 1 (1)
Allergy-Other (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hemoglobinuria (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vasovagal episode (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vision-blurred vision (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyramidal tract dysfunction (e.g., increased tone, hyperreflexia, positive Babinski, decreased fine (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rigors/chills (General disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Lymphopenia (Investigations) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Laryngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anorexia (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Arrhythmia-Other (Cardiac disorders) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Ataxia (incoordination) (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bilirubin (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chest pain (non-cardiac and non-pleuritic) (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Constitutional symptoms-Other (General disorders) | 0 (0) | 2 (4) | 0 (0) | 0 (0)
Fever (in absence of neutropenia where neutropenia is defined as AGC<1.0x109)L (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dysuria (painful urination) (Renal and urinary disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Extrapyramidal/involuntary movement/restlessness (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
A total of 159 participants were accrued beginning in March 2000 until January 2005. Accrual rates were less than anticipated and the study was closed to further entry by the Independent Data Safety and Monitoring Board for the NCI CCR.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2009-05-20): https://cdn.clinicaltrials.gov/large-docs/35/NCT00004635/Prot_000.pdf
  • Informed Consent Form (2005-04-28): https://cdn.clinicaltrials.gov/large-docs/35/NCT00004635/ICF_001.pdf